CLINICAL TRIAL: NCT01433952
Title: Pharmacokinetics of High Dose Oral Thiamine
Brief Title: Pharmacokinetics of Oral Thiamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 132653
Record Dates: First submitted 2011-09-07; First posted 2011-09-14 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Pharmacokinetics in Healthy Subjects
MeSH Terms: interventions — Thiamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0 mg Thiamine (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- 100 mg Thiamine (Experimental)
  Interventions: Dietary Supplement: Thiamine
- 500 mg Thiamine (Experimental)
  Interventions: Dietary Supplement: Thiamine
- 1500 mg Thiamine (Experimental)
  Interventions: Dietary Supplement: Thiamine

INTERVENTIONS:
Dietary Supplement: Thiamine — Vitamin B1
  Arms: 100 mg Thiamine; 1500 mg Thiamine; 500 mg Thiamine
Dietary Supplement: Placebo — Placebo
  Arms: 0 mg Thiamine

SUMMARY:
Elevated levels of thiamine may increase cellular energy metabolism by increasing the activity of pyruvate dehydrogenase complex. This has been hypothesized to have a beneficial affect in patients with several diseases including sepsis, heart failure, and diabetes. There is limited data on the pharmacokinetics of supraphysiologic doses of oral thiamine.

The aims of this study are to:

* Calculate the plasma and whole blood pharmacokinetics of supraphysiologic doses of oral thiamine in healthy volunteers;
* Compare the different thiamine doses on the pharmacokinetic variables using repeated measures ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55

Exclusion Criteria:

* Non dietary thiamine supplement within two weeks of the start of the study or during the study
* History of thiamine deficiency
* Anemia (Hgb<10)
* History of gastrointestinal absorption disorders
* Taking prescription or over-the-counter medication
* Pregnant or breast feeding a child
* Alcohol and or drug abuse
* Smoker

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) for whole blood | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 hours post-dose
Area Under the Curve (AUC) for plasma | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Howard Smithline, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States